CLINICAL TRIAL: NCT03061747
Title: Italian Multi-centre Observational Registry on Patients With impLANTable Devices Remotely monitorED
Brief Title: Multi-centre Observational Registry on Patients With Implantable Devices Remotely Monitored
Acronym: IMPLANTED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Responsible Party: Sponsor
Other Study IDs: IMPLANTED
Record Dates: First submitted 2017-02-18; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Defibrillators, Implantable; Heart Failure With Reduced Ejection Fraction; Arrythmia; Pacemaker
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Assesment of outcome of implantable device patients — Evaluation during follow-up of the occurrence of atrial arrhythmias, hospitalizations, and of death.

SUMMARY:
Multicentric, observational, retrospective registry including patients underwent implantable device implantation (pacemaker or ICD) for any indication in the period from 2009 to 2016, followed by remote monitoring. The aims of the registry are to evaluate the occurrence of atrial arrhythmias, of hospitalizations, and the mortality during a long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* ICD of pacemaker implantation fo any indication
* Followed by remote monitoring
* Age >18 years

Exclusion Criteria:

* life expectancy of less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients underwent ICD or pacemaker implantation from January 2009 to September 2016 for any indication and followed by remote monitoring at enrolling hospitals
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-04-15 (Estimated); Study Completion 2017-04-30 (Estimated)

PRIMARY OUTCOMES:
Death for any cause | an average of 2 years

SECONDARY OUTCOMES:
Atrial arrhythmias | an average of 2 years
Hospitalizations for any cause | an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Palmisano, MD, Principal Investigator — Card. G. Panico Hospital - Tricase - Italy
Locations (6):
- Italy (6):
  - Policlinico S.Orsola-Malpighi, Bologna, Bologna
  - AO Pugliese-Ciaccio, Catanzaro, Catanzaro
  - Dell'Era Gabriele, Novara, Novara
  - University Hospital "Umberto I - Lancisi - Salesi", Ancona
  - Vito Fazzi Hospital, Lecce
  - Monaldi Hospital, Napoli